CLINICAL TRIAL: NCT07276542
Title: PHANTOM LIMB PAIN KETAMINE TREATMENT STUDY
Brief Title: Clinical Trial Exploring the Outpatient Treatment of Phantom Limb Pain With Ketamine Administration in a Six Month Study With a Minimum Remission Period of 7 Days Between Treatment Session. 25-30 Subjects With an Ongoing History of Significant PLP.--FDA and IRB Approved.
Acronym: PLP
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Ketamine Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRF-PLP; IND 175124 (Other: FDA)
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Phantom Limb Syndrome With Pain
Keywords: Phantom Limb Pain, PLP. ketamine, ketamine and pain, ketamine assisted psychotherapy
MeSH Terms: conditions — Phantom Limb; Pain

STUDY DESIGN:
Intervention Model Description: Provision of IM ketamine in a protocol with minimal time for response of 7 days and assessment of need for treatment over six months' time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PLP Ketamine Intervention (Experimental)
  Interventions: Drug: IM ketamine in dose finding and then continuation

INTERVENTIONS:
Drug: IM ketamine in dose finding and then continuation — Intermittent ketamine treatment based on response

SUMMARY:
An anecdotal report with administration of ketamine in a non-clinical setting providing and sustained remission of symptoms after 6 years has furthered the interest in ascertaining if ketamine might indeed be a successful intervention. (See Wolfson and Barocchi).

Ketamine has shown benefit in a variety of pain and neurological disorders. Its exploration for these continues and there appears to be an expanding use of ketamine for difficult to treat syndromes. Phantom limb pain occurs in over 50% of amputees, tends to be immediate in onset, but may occur at a later time. It is often excruciating, with a high frequency of episodes that tend to diminish with time-- variably. Its treatment is reliant on opioids and other pain medications usually with limited results. Acupuncture has been minimally explored with no clear results. Our study aims at clarifying ketamine's status for this particular disorder.

This is an off-label use of RS ketamine for clinical purposes. Each subject of the 25-30 enrolled in the study will have up to 16 ketamine sessions over six months time, Subjects will be continued in the study if the partial or complete remission period is seven days or more, If less, subjects will be considered to have not adequately responded to the protocol's provision of IM ketamine. Dosage of ketamine will be determined in the initial session with a dosage escalation protocol with an upper limit of 120mg--that limit not to be exceeded for the duration of each subject's participation in the study.. The time for a succeeding session of ketamine is variable depending on response and therefore the duration of the remission--not to be less than 7 days as the minimum consideration for a response, Subjects will receive support throughout their sessions and these will be conducted with integration following the medication, much as in the ketamine assisted psychotherapy model practiced by us as clinicians.

As PLP has its emotional impact as well as its complex pain presentation, these parameters will be followed with a variety of assessment tools. The nature of each subjects PLP syndrome will be analyzed in detail as well as the particularity of responses to the elements of the syndrome..

ELIGIBILITY:
Inclusion Criteria:

* Presence of phantom limb pain at the time of administration of ketamine.
* Willingness to participate in the study and follow-up over a year long period.
* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* If female, must have a negative pregnancy test at Screening and any subsequent administration of ketamine. Sexually active females and male partners must be using adequate birth control measures during the duration of the study when ketamine will be administered and for one week after the last administration of ketamine.
* Patient agrees to withhold alcohol, marijuana, nicotine products, and any other intoxicants for at least 24 hours
* Normotensive-defined as Abnormal VS, after 5 minutes supine rest at Screening or on Day -1, defined as any of the following:

Systolic BP> 150 mmHg.

* Diastolic BP> 105 mmHg.
* HR <50 or >110 bpm.

  * Not on Medications that would blunt ketamine's effects
  * 18-65
  * No prior history of treatment with ketamine for PLP.

Exclusion Criteria:

Exclusion Criteria

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study.
* Vulnerable persons are Excluded from the study. This includes subjects with known psychotic illness, mania, significant neurologic disorders, elevated intraocular and or intracranial pressures
* Exclusion of subjects with abnormal baseline hepatic and renal lab tests.
* Exclusion of subjects with cardiovascular disease, arrythmias, or abnormal EKGs.
* The presence of any medication that might cause an adverse reaction with ketamine.
* The Ketalar Label as cited by FDA includes Drug Interactions particular to anesthesia and the use of IV boluses at far higher dosages than those used in our study. In Review of these:

Theophylline Or Aminophyline --Excluded

* Sympathomimetics And Vasopressin-Excluded
* Benzodiazepines-PLP patients may be on benzodiazepines or other anxiolytic medications, Subjects will be asked to suspend daytime use of these whenever possible recognizing that anxiety is an often present symptom within the PLP complex. Recognition of a possible increase in sedation due to the concomitant presence of a benzodiazepine with ketamine may lead to a lowering of the ketamine dosage. Nighttime use of a benzodiazepine for treatment of insomnia will not be discontinued unless the dosage is high and considered to have a sedating effect on the degree of ketamine's sedation the next day. The length of time between nighttime use and administration of ketamine during the day should diminish the effects of the nighttime medication.
* Opioid Analgesics -PLP subjects most likely will have been or will be receiving opiates for pain relief, Concomitant use of ketamine and opiates in outpatient settings for analgesia is a common and accepted practice. Withdrawing opiates for ketamine administered in subanesthetic doses is not appropriate. In several studies ketamine has been shown to reduce the amount of opioids needed for analgesia, It is the hope of this study that successful treatment with ketamine will enable reduction or cessation of opioid use, In our vast clinical experience, we have treated with ketamine at subanesthetic doses patients on opiates without adverse effects.
* Subjects on long-acting opioids such as methadone or extended-release opioids are excluded.
* Subjects with opioid use 50 mg/day MME (morphine milliequivalents) within 1 week of initial ketamine administration are excluded.
* Subjects with +UDS (urine drug screen) for ketamine, cocaine, methamphetamine, PCP, or other substances of abuse are excluded.
* Subjects who have used THC may be enrolled but must have abstained from THC for at least 3 days prior to each ketamine session

Concomitant medications:

* Oral IR (immediate release) opioid mu agonists up to 50 mg/day MME (morphine milliequivalents) are allowed (e.g., hydromorphone, oxycodone, morphine, and hydrocodone).
* No increases of any opioids or other concomitant medications, or addition of new medications or therapies for PLP will be allowed during the study.
* All concomitant medications, including type and amount, will be recorded by study participants in their daily diaries and reviewed by study staff before each treatment session and any scheduled telephone calls.
* Participants will not receive opioids 4 hours before or after ketamine administration.
* Laboratory assessments: Subjects with abnormal baseline hepatic or renal lab tests are to be excluded. In addition, obtain the following laboratory tests at the following times: CBC, hepatic and renal labs at 3 months and 6 months. Follow-up abnormal laboratory values.
* Or Other CNS Depressants-gabapentin may well be prescribed for patients with PLP as is true for pregabalin, Whenever possible subjects will be asked to withhold these for at least 4 hours prior and not resume for at least 4 hours after the last administration of ketamine. This is consistent with two half-lives of ketamine
* Alcohol-Daily use exceeding 2 US Standard drinks. No alcohol use in 24 hours preceding a ketamine session.
* Stimulants-Subjects will be asked to withhold stimulants for 5-12 hours prior to administration of ketamine depending on the duration of action of the particular preparation and not resume until the next day after treatment.

Inclusion Criteria:

-

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
McGill Pain Questionnaire SF-MPQ-2 | 6 months per subject with a 12 month follow-up
  A complex assassement measure for complex pain presentations

CONTACTS AND LOCATIONS:
Locations (1):
- Ketamine Research Foundation, San Anselmo, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Outcome data for each participant

REFERENCES:
- See also: Parent non-profit organization for study--Sponsor — http://www.ketamineresearchfoundation.org